CLINICAL TRIAL: NCT03908073
Title: Electrical Vagal Nerve Stimulation in Ulcerative Colitis - a Double Blind Placebo - Controlled Study of Transcutaneous Vagal Nerve Stimulation in Ulcerative Colitis
Brief Title: Electrical Vagal Nerve Stimulation in Ulcerative Colitis
Acronym: EVASION-UC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 18/LO/1693
Record Dates: First submitted 2019-02-22; First posted 2019-04-09 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2019-01

CONDITIONS: Ulcerative Colitis; Vagal Nerve Stimulation; Transcutaneous Vagal Nerve Stimulation
Keywords: Ulcerative Colitis; Vagal Nerve Stimulation; Transcutaneous Vagal Nerve Stimulation; Cytokines; LPS stimulated cytokine production
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: Proof of concept prospective randomized double-blind crossover study evaluating the use of transcutaneous vagal nerve stimulation in a model of acute psychological stress in participants with quiescent Ulcerative colitis
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active transcutaneous vagal nerve stimulation (Active Comparator): The participant will be taught how to use the device and administer doses in our laboratory and independently at home over a period of 24 hours.
  Interventions: Device: Transcutaneous vagal nerve stimulation
- Sham transcutaneous vagal nerve stimulation (Placebo Comparator): The participant will be taught how to use the device and administer doses in our laboratory and independently at home over a period of 24 hours.
  Interventions: Device: Transcutaneous vagal nerve stimulation

INTERVENTIONS:
Device: Transcutaneous vagal nerve stimulation — The use of a transcutaneous vagal nerve stimulator by the participant

SUMMARY:
There are approximately 2.5-3 million patients with inflammatory bowel disease (IBD) across Europe, with associated healthcare costs of €4.6-5.6 billion per annum (1). IBD is associated with a significant reduction in quality of life. Treatments directed towards modifying the inflammatory response, such as anti-tumour necrosis factor-alpha (TNF-α) agents, are expensive, can necessitate admission to hospital for their administration and can be associated with side effects (2 3). Thus, the development of a novel non-pharmacological anti-inflammatory intervention, such as electrical vagal nerve stimulation, is warranted.

This is a proof of concept study which aims to investigate whether transcutaneous vagal nerve stimulation is effective at reducing stress induced inflammatory cytokine levels in patients with quiescent ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between 18 and 76 years of age (inclusive).
* Has a clinical diagnosis of UC at least 3 months before screening according to accepted international guidelines.
* Quiescent disease. Disease activity will be assessed using the validated partial Mayo score and faecal calprotectin of <4 and <250 μg/g (18) respectively, scored within 3 months of entry into the study. Faecal calprotectin <250 μg/g within 2 weeks before study entry to confirm that there has been no change in activity status.
* Stable medications regimen for 3 months prior to entry into the study, defined as no additions to UC treatment or dosage escalations.
* Patient is willing and able to participate in the study for the required duration, can understand and is willing to sign the ICF and agrees to undergo all protocol-related tests and procedures.
* Patient has a BMI between 18 and 35 kg/m2 inclusive.

Exclusion Criteria:

* Has severe extensive colitis and is at imminent risk of colectomy.
* Presence of a stoma or history of a fistula.
* Currently taking any topical or oral corticosteroids.
* Currently taking any anti-TNF therapy, azathioprine, 5-mercaptopurine or methotrexate.
* Is pregnant, lactating or thinking of becoming pregnant during the study period, or of childbearing years and is unwilling to use and accepted form of birth control.

(Female patients of child-bearing potential must have a negative urine pregnancy test at Screening/pre-dose on Day 1 of the study, excluding female patients of non-child bearing potential who are surgically sterile or post-menopausal. [To be considered post-menopausal female patients must be without menses for 12 consecutive months before screening].)

* Patient has unstable acute illness or exacerbation or an unstable chronic illness or chronic disease (other than UC) that may affect assessments for this study as determined by previous physical examination, medical history, vital signs, ECG, and laboratory (serum biochemistry, haematology, urinalysis) assessments. (Note: Non-fasting elevations of cholesterol and triglycerides are not considered clinically significant.)
* Patient with medical history of hepatitis B, hepatitis C or human immunodeficiency virus (HIV) infection
* Has known or suspected severe cardiac disease (e.g., symptomatic coronary artery disease, prior myocardial infarction, congestive heart failure (CHF);
* Has known or suspected cerebrovascular disease (e.g. prior stroke or transient ischemic attack, symptomatic carotid artery disease, prior carotid endarterectomy or other vascular neck surgery);
* Has a clinically significant abnormal screening Electrocardiogram (ECG) e.g. second and third degree heart block, prolonged QT interval, atrial fibrillation, atrial flutter, history of ventricular tachycardia or ventricular fibrillation, or clinically significant premature ventricular contraction);
* Has had a cervical vagotomy;
* Has uncontrolled high blood pressure (systolic >160, diastolic >100 after 3 repeated measurements within 24 hours);
* Is currently implanted with an electrical and/or neurostimulator device (e.g.. cardiac pacemaker or defibrillator, vagal neurostimulator, deep brain stimulator, spinal stimulator, bone growth stimulator, cochlear implant, sphenopalatine ganglion stimulator or occipital nerve stimulator);
* Has been implanted with metal cervical spine hardware or has a metallic implant near the gammaCore® stimulation site;
* Has a history of syncope (within last two years);
* Has a history of seizures (within last five years);
* Has a known history or suspected history of substance abuse or addiction (within last five years);
* Has previously used the gammaCore® device.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
The effect of active transcutaneous vagal nerve stimulation on LPS stimulated TNF-α production in comparison to sham after the stress protocol | 1 year
  Whole blood taken from the participants is stimulated with LPS. The concentration of TNF-α will be measured using the ELISA technique. TNF-α level of intervention versus sham is the primary outcome measure.

SECONDARY OUTCOMES:
The effect of active transcutaneous vagal nerve stimulation compared to sham on LPS stimulated TNF-α production without the stress protocol | 1 year
  Whole blood taken from the participants is stimulated with LPS. The concentration of TNF-α will be measured using the ELISA technique. TNF-α level of intervention versus sham without the stress protocol is a secondary measure.
Cardiac vagal tone at baseline visits 1 and 2 and post stress protocol | 1 year
  Cadriac vagal tone and autonomic nervous system monitoring is performed in our laboratory using a specialised device called 'powerlab'.
  It is able to convert ECG data into autonomic parameters, including vagal tone, which the investigators can then use as an outcome measure.
The effect of active transcutaneous vagal nerve stimulation compared to sham on LPS stimulated Il6 and Il10 production with and without the stress protocol | 1 year
  Whole blood taken from the participants is stimulated with LPS. The concentration of IL6 and IL10 will be measured using the ELISA technique. IL6 and IL10 level of intervention versus sham without the stress protocol is a secondary measure.

CONTACTS AND LOCATIONS:
Locations (1):
- Tamara Mogilevski, London, Select One, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mogilevski T, Hardy MY, Takahashi K, Smith R, Nguyen AL, Farmer A, Lindsay JO, Tye-Din JA, Aziz Q, Gibson PR. Effects of Stress, Vagal Nerve Stimulation and Disease Activity on Circulating Cytokines, Quantified by an Ultrasensitive Technique, in Ulcerative Colitis: A Pilot Study. JGH Open. 2025 Jun 28;9(7):e70206. doi: 10.1002/jgh3.70206. eCollection 2025 Jul. PMID 40584280